CLINICAL TRIAL: NCT03123315
Title: Optimization of Parameters for Ureterolysis During Minimally Invasive Hysterectomy; Determining Variation in Ureter Position and Degree of Thermal Spread
Brief Title: Optimization of Ureterolysis During Hysterectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: per PI request
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE11815
Record Dates: First submitted 2017-04-14; First posted 2017-04-21 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Hysterectomy
Keywords: hysterectomy; ureter

STUDY DESIGN:
Intervention Model Description: Single-Center Prospective Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cook Bush DL™ Ureteral Illuminating Catheter (Experimental): As part of this study an additional tool will be used during the hysterectomy. This tool is called a Cook Bush DL™ Ureteral Illuminating Catheter, which is a lighted ureteral stent. This is a very thin tube that goes into the ureter. A urologist, who is an expert at placing these devices, will insert a stent into each ureter during surgery. The lighted stents will help effectively find the ureters and keep track of them during the surgery. This same procedure is already being done in many other forms of abdominal surgery to help find the ureter. The stents will be removed before the surgery is complete and treatment will not differ in any other way.
  Interventions: Device: Ureteral Illuminating Catheter

INTERVENTIONS:
Device: Ureteral Illuminating Catheter — This is a very thin tube that goes into a ureter to more effectively find and track the ureter during surgeries
  Other Names: ureteral stent

SUMMARY:
The purpose of this study is to improve the safety of surgery to remove a uterus (a hysterectomy) by better understanding where a patient's ureters lie.

DETAILED DESCRIPTION:
Objectives:

Primary: (While uterus is under tension)

* To determine the shortest distance from the ureter to the uterine vessels.
* To determine the distances from the ureter to the gonadal vessels in infundibulo-pelvic (IP) at the pelvic sidewall. This will be defined at the distance from the IP ligament at the level of the pelvic sidewall to the point on the ureter directly below these vessels
* To determine the distances from the ureter to the gonadal vessels in the infundibulo-pelvic (IP) ligament at the point where the gonadal vessels enter in to the ovary. This will be defined as the distance from where the vessels in the IP enter the ovary to the point on the ureter directly below this.

Secondary

* To determine thermal spread from the Ligasure, and Harmonic device using H&E and Movat staining.
* To determine the burst pressure of segments of IP ligament that have undergone Ligasure or Harmonic electrosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing minimally invasive surgery (MIS) hysterectomy with Bilateral Salpingo Oophorectomy (BSO) for either a benign or malignant condition.
* Performance Status of 0-1
* Must have the ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* History of radical pelvic surgery.
* History of stage IV-V uterine prolapse or hysteropexy
* History of prior ureteral injury or retroperitoneal dissection
* Known hydronephrosis.
* Known congenital genitourinary or gynaecologic anomaly
* Any known obstructing mass along any portion of the pelvic ureter
* Known American Society for Reproductive Medicine (ASRM) stage III/IV endometriosis (obliteration of the cul-de-sac)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Distance from the ureter to the uterine vessels | Cross-sectional measurement at time of surgery
  To determine the shortest distance from the ureter to the uterine vessels to show the variation of ureteral position to the uterine and gonadal vessels during total laparoscopic hysterectomy prior to and following opening the retroperitoneum. Lighted ureteral stents will be placed cystoscopically. This will be done to clearly delineate the ureter and facilitate measuring the ureter to the infundibulopelvic (IP) and ureter to uterine vessel distances.
The distance from the ureter to the right gonadal vessel at the pelvic sidewall | Cross-sectional measurement at time of surgery
  To determine the average distance from the ureter to the right gonadal vessel in infundibulo-pelvic (IP) at the pelvic sidewall. This is to show the variation of ureteral position to the uterine and gonadal vessels during total laparoscopic hysterectomy prior to and following opening the retroperitoneum. Lighted ureteral stents will be placed cystoscopically. This will be done to clearly delineate the ureter and facilitate measuring the ureter to the infundibulopelvic (IP) and ureter to uterine vessel distances.
The distance from the ureter to the left gonadal vessel at the pelvic sidewall | Cross-sectional measurement at time of surgery
  To determine the distance from the ureter to the left gonadal vessel in infundibulo-pelvic (IP) at the pelvic sidewall. This is to show the variation of ureteral position to the uterine and gonadal vessels during total laparoscopic hysterectomy prior to and following opening the retroperitoneum. Lighted ureteral stents will be placed cystoscopically. This will be done to clearly delineate the ureter and facilitate measuring the ureter to the infundibulopelvic (IP) and ureter to uterine vessel distances.
The distance from the ureter to the right gonadal vessel where the gonadal vessel enter in to the ovary | Cross-sectional measurement at time of surgery
  To determine the distance from the ureter to the right gonadal vessel in the infundibulo-pelvic (IP) ligament at the point where the gonadal vessels enter in to the ovary. This is to show the variation of ureteral position to the uterine and gonadal vessels during total laparoscopic hysterectomy prior to and following opening the retroperitoneum. Lighted ureteral stents will be placed cystoscopically. This will be done to clearly delineate the ureter and facilitate measuring the ureter to the infundibulopelvic (IP) and ureter to uterine vessel distances.
The distance from the ureter to the left gonadal vessel where the gonadal vessel enter in to the ovary | Cross-sectional measurement at time of surgery
  To determine the distance from the ureter to the left gonadal vessel in the infundibulo-pelvic (IP) ligament at the point where the gonadal vessels enter in to the ovary. This is to show the variation of ureteral position to the uterine and gonadal vessels during total laparoscopic hysterectomy prior to and following opening the retroperitoneum. Lighted ureteral stents will be placed cystoscopically. This will be done to clearly delineate the ureter and facilitate measuring the ureter to the infundibulopelvic (IP) and ureter to uterine vessel distances.

SECONDARY OUTCOMES:
To determine the burst pressure of infundibulopelvic (IP) ligament which had Ligasure electrosurgery | Cross-sectional measurement at time of surgery
  To determine the burst pressure of segments of IP ligament that have undergone Ligasure electrosurgery. The Ligasure electrosurgery cuts and seals the tissue during surgery. The burst pressure gives a measure of how well the tissue is sealed.
To determine the burst pressure of infundibulopelvic ligament which had Harmonic electrosurgery | Cross-sectional measurement at time of surgery
  To determine the burst pressure of segments of IP ligament that have undergone Harmonic electrosurgery. The Harmonic electrosurgery cuts and seals the tissue during surgery. The burst pressure gives a measure of how well the tissue is sealed.

OTHER OUTCOMES:
To determine thermal spread from a Ligasure to show the | Cross-sectional measurement immediately after surgery
  Thermal spread is the dispersal of heat into surrounding tissue during electrosurgeries, causing damage to the tissue.In order to measure thermal spread, the gonadal vessels will be harvested after the specimen (uterus, tubes, ovaries and cervix) has been removed from the patient
To determine thermal spread from a Harmonic device | Cross-sectional measurement immediately after surgery
  Thermal spread is the dispersal of heat into surrounding tissue during electrosurgeries, causing damage to the tissue. In order to measure thermal spread, the gonadal vessels will be harvested after the specimen (uterus, tubes, ovaries and cervix) has been removed from the patient

CONTACTS AND LOCATIONS:
Overall Officials: Robert Debernardo, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center